CLINICAL TRIAL: NCT02100293
Title: Effects of Magnesium Sulfate on Onset and Duration of Low Dose Rocuronium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1307/209-006
Record Dates: First submitted 2013-12-11; First posted 2014-03-31 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2015-07

CONDITIONS: Observation of Neuromuscular Block; Intubation Condition; Surgical Condition
Keywords: magnesium sulfate, rocuronium
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard dose rocuronium group (Active Comparator): pretreatment of saline 100ml and rocuronium 0.6 mg/kg
  Interventions: Drug: saline
- low dose rocuronium group (Active Comparator): pretreatment of saline 100ml and rocuronium 0.45 mg/kg
  Interventions: Drug: saline
- low dose rocuronium plus magnesium group (Active Comparator): pretreatment of magnesium sulfate 30 mg/kg and rocuronium 0.45 mg/kg
  Interventions: Drug: magnesium sulfate 30 mg/kg

INTERVENTIONS:
Drug: magnesium sulfate 30 mg/kg — Patients in each group received the magnesium sulfate 30 mg/kg for 2 min in 0.9% normal saline (total volume 100 ml) intravenously for 5 min before induction of anesthesia
  Arms: low dose rocuronium plus magnesium group
Drug: saline — Patients in each group received 0.9% normal saline (total volume 100 ml) alone intravenously for 5 min before induction of anesthesia
  Arms: low dose rocuronium group; standard dose rocuronium group

SUMMARY:
This study aims to evaluate effects of magnesium sulfate on onset and duration of low dose rocuronium, intubation condition and surgical condition.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 yr American Society of Anesthesiologists physical status 1 or 2, BMI of 20-24.9 kg/m2 scheduled for elective laryngeal microsurgery

Exclusion Criteria:

* severe respiratory or cardiac disease hepatic or renal function impairment neuromuscular disease on medications affecting neuromuscular function with known allergy to the drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
onset time of rocuronium | from injection of rocuronium to T1 suppression more than 95% up to 10 minutes
  from injection of rocuronium to T1 suppression more than 95% up to 10 minutes

SECONDARY OUTCOMES:
maximal suppression time and duration of rocuronium | time from the injection of rocuronium to T1 maximal suppression time and reversal of T1 25% up to 1 hours

OTHER OUTCOMES:
intubation condition | intubation condition during induction of anesthesia up to 10 minutes
  We scored intubation condition on the basis of 4 items, laryngoscopy, vocal cord position, moving of limbs, and coughing.
surgical condition | intraoperative surgical condition
  to score a surgical condition according to 7 point likers scale
postoperative sore throat | postoperative sore throat up to 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hwan Do, Principal Investigator — Seoul National Univ. Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospita, Seongnam-si, Gyeonggi-do, South Korea